CLINICAL TRIAL: NCT05218577
Title: The Effect of High Selenium Functional Food and Selenium Supplement on Developmental Level in Autism Spectrum Disorder
Brief Title: The Effect of High Selenium Functional Food and Selenium Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neny Triana (Other)
Responsible Party: Sponsor-Investigator, Neny Triana, STIKES Karya Husada Kediri, Karya Husada Sshool Health Science
Organization: Karya Husada Sshool Health Science (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neny Triana
Record Dates: First submitted 2022-01-30; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The Intervention group were given HSFF and selenium suplemen, and control group was given placebo.
Who Masked: Participant, Investigator
Masking Description: participant did'n know what they had got. the investigator did'n know group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSFF group (Experimental): the group was given high selenium funtion selenium for 3 months
  Interventions: Other: high selenium functional food
- Selenium suplemen group (Experimental): the group was given selenium suplemen
  Interventions: Dietary Supplement: selenium supplement
- Control group (Placebo Comparator): the group was given placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: high selenium functional food — HSFF was made from the liver of the cow, that participant could eat HSFF direcly.
  Other Names: HSFF
  Arms: HSFF group
Dietary Supplement: selenium supplement — 20 microgram/day selenium suppplement powder.
  Arms: Selenium suplemen group
Other: Placebo — the placebo mocaf powder
  Arms: Control group

SUMMARY:
The prevalence of ASD is increasing every year. Report data from the Center for Diseases Control and Prevention (CDC) 1: 68 in 2016 means that out of 68 children, there is 1 child with ASD, while in 2017 it increased by 1: 36, meaning that out of 36 children there is 1 child with ASD1. ASD in men is 4 times greater than in women. This study used Randomized Controlled Clinical Trials (RCT), double blind, 65 research subjects randomized to provide intervention for 3 months in group 1 (n = 22) processed beef liver high in selenium, group 2 (n = 22) supplemented with selenium, group 2 (n = 22) supplemented with selenium, group 1 (n = 22) 3 (n=21) control group. Outcome of ATEC score measurement in the three groups. Major hypothesis There is a difference in the comparison of giving high selenium functional food (HSFF) with selenium supplements to decreasing ATEC scores in Autism Spectrum Disorder (ASD) children, increasing levels of the enzyme glutathione peroxidase (GPx), and decreasing IL-β, IL-6 and TNF-α . Minor Hypothesis. a. There was a decrease in the ATEC score of ASD children in the intervention group of processed beef liver high in selenium, selenium supplementation compared to the control group b. The difference in the increase in GPx enzyme levels in the intervention group processed beef liver high in selenium, selenium supplementation compared to the control group in ASD children. c. Differences in decreased levels of IL-1β in the intervention group processed beef liver high in selenium, selenium supplementation compared to the control group with ASD.d. Differences in decreased levels of IL-6 in the intervention group processed high-selenium beef liver, selenium supplementation compared to the control group with ASD children. e. Differences in decreased levels of TNF- in the intervention group processed beef liver high in selenium, selenium supplementation compared to the control group with ASD children. Participants were randomized into three groups: Intervention group 1 high selenium functional food (n=22), Intervention 2 selenium supplement and group 3 control (n=21).

DETAILED DESCRIPTION:
Introduction:

Autism Spectrum Disorder (ASD) is a developmental disorder, which is characterized by two symptoms, namely, barriers to communication/social interaction and restrictive/repetitive behavior. Knowing children with ASD, parents reported their children at the age of 18 months with verbal and non-verbal speech delays compared to children their age. To find out as early as possible children with ASD, it is necessary to be screened at the age of 18 and 24 months, before a diagnosis of ASD is made based on the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders-5), this is to conduct early intensive intervention in improving the disorder. its development. The prevalence of ASD is increasing every year. Report data from the Center for Diseases Control and Prevention (CDC) 1: 68 in 2016 means that out of 68 children, there is 1 child with ASD, while in 2017 it increased by 1: 36, meaning that out of 36 children there is 1 child with ASD1. ASD in men is 4 times greater than in women.

The causes of ASD are non-genetic and genetic. Non genetic include, neuroinflammation and neuroimmunity, digestive disorders, neuropathology, heavy metal poisoning. Inflammation of the innervation of children with ASD causes the production of pro-inflammatory cytokines to increase. Cytokines that play a role in ASD innervation are IL-1 , IL-6 and TNF-α. These cytokines can cross the blood-brain barrier, thereby influencing behavior in ASD. Children with ASD also experience bacterial abnormalities in their stools. Based on the results of the study of bacterial cultures in the feces of children with ASD, significant Bifidobacterium, Escherichia coli, Lactobacillus, and Enterococcus bacteria were found. This increase in faecal flora indicates intestinal inflammation in ASD children, this causes the blood brain barrier to be disrupted, because the intestinal function that provides nutrients to neurons is not optimal, thus affecting the work of the nervous system as a trigger for neuroinflammation. Heavy metal poisoning, in ASD there was an increase in the concentration of Hg in the hair, and there was a significant relationship between lead content in ASD hair and the development of verbal communication (p= 0.020). Genetic factors, ± 15% ASD It is estimated that 37%-90% of siblings with ASD twins will be at risk of developing ASD in their siblings.

Interprofessional ASD handling involves inter-professional collaboration pediatricians, psychologists, nurses, medical rehabilitation, and nutritionists working as a team to help families with ASD children. Early treatment before the age of 3 years, highly recommended. The goal of ASD treatment is to maximize the child's independence and quality of life by minimizing the symptoms of ASD development. Treatment with Complementary and Alternative Medicine (CAM) is used for the prevention, cure and promotion of ASD. CAM is divided into biological therapies including casein free, gluten free, sugar free (CFGFSF) dietary interventions, supplements, and non-biological, including social therapy, hearing integration training, sensory integration therapy, drama therapy, dance therapy, acupuncture, massage therapy, yoga and animal therapy.

One of the treatments for CAM with biologic therapy in ASD is selenium supplementation, where selenium is essential for specific, non-specific, and antioxidant immune responses. Selenium given to ASD, is a selenoprotein element as an essential component of the enzyme glutathione peroxidase (GPx). GPx acts to reduce hydrogen peroxide (H₂O₂) to water (H2O), improve neuronal degeneration and release reactive oxygen species (ROS) due to oxidative stress. Selenium as an antioxidant compound, is a compound that works by donating one electron or giving electrons (electron donors) to compounds that are oxidant, so that the activity of these oxidant compounds can be inhibited.

Formulation of the problem:

Can administration of high selenium functional food (HSFF) reduce ATEC scores in developing ASD children, increase GPx, decrease IL-1 , IL-6, and TNF- compared to selenium supplements

Research purposes:

Proving the comparison of giving high selenium functional food (HSFF) with supplemental selenium (SS) on the clinical development of ASD children, can decreased ATEC score, increased GPx, decreased IL-1 , IL-6, and TNF-α.

Research Hypothesis:

There is a difference in the comparison of giving high selenium functional food (HSFF) with selenium supplements to decreasing ATEC scores in children with Autism Spectrum Disorder (ASD), increasing levels of the enzyme glutathione peroxidase (GPx), and decreasing IL-β, IL-6 and TNF-α.

Benefits of research:

Provides academic benefits in improving pediatric nursing knowledge, the immune system IL-1β, IL-6, and TNF-α and GPx antioxidants related to high-slenium beef liver preparations and selenium supplements in the development of ASD children.

Research methods:

A true experimental study with a randomized controlled group pre-post test design. The research subjects were ASD boys and girls (n=65), divided into 3 groups, 22 subjects were given processed beef liver high in selenium, 22 subjects were supplemented with selenium, 21 subjects were controls. The characteristics of the research subjects included age, gender, first diagnosed with ASD, knowledge of diet and doctor's therapy. Each group was assessed for development by ATEC scores, levels of GPx, IL-1β, IL-6 and TNF-α before and after the intervention. The intervention group 1 was given processed beef liver with high selenium, the intervention group 2 was given selenium supplementation and group 3 as a control was given mocaf flour for 3 months.

The normality test of the data distribution was carried out by Kolmogorov-Smirnov, to determine the results before and after the intervention with the paired, unpaired t-parametric test and One Way Anova and the non-parametric Chi-Square test, Kruskal Wallis.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with ASD by a pediatrician, based on DSM-5
2. ASD children aged 2-6 years.
3. ASD children receiving medical and non-medical therapy.

Exclusion Criteria:

1. ASD children who were not at the study site.
2. Children with ASD are accompanied by severe congenital abnormalities.

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
The change of Developmental level | Baseline and 3 month after the intervention
  Developmental level was measured by Autism Treatment Evaluation Cheecklist (ATEC)

SECONDARY OUTCOMES:
The change of GPx level | Baseline and 3 month after the intervention
  Gluthation peroxidase is antioxidant that measured in the laboratory using elisa method
The change of IL-1 betha level | Baseline and 3 month after the intervention
  IL-1 Betha is pro inflamation that measured in the laboratory using elisa method
The change of IL-6 level | Baseline and 3 month after the intervention
  IL-6 is pro inflamation that measured in the laboratory using elisa method
The change of TNF-Alpha level | Baseline and 3 month after the intervention
  TNF-Alpha is pro inflamation that measured in the laboratory using elisa method

CONTACTS AND LOCATIONS:
Overall Officials: Neny Triana, Principal Investigator — STIKES Karya Husada Kediri
Locations (1):
- Neny Triana, Kediri, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
I did'd have a plan share the date

REFERENCES:
- [Result] Brondino N, Fusar-Poli L, Rocchetti M, Provenzani U, Barale F, Politi P. Complementary and Alternative Therapies for Autism Spectrum Disorder. Evid Based Complement Alternat Med. 2015;2015:258589. doi: 10.1155/2015/258589. Epub 2015 May 7. PMID 26064157
- [Result] Sharma SR, Gonda X, Tarazi FI. Autism Spectrum Disorder: Classification, diagnosis and therapy. Pharmacol Ther. 2018 Oct;190:91-104. doi: 10.1016/j.pharmthera.2018.05.007. Epub 2018 May 12. PMID 29763648
- [Result] Lange KW, Hauser J, Reissmann A. Gluten-free and casein-free diets in the therapy of autism. Curr Opin Clin Nutr Metab Care. 2015 Nov;18(6):572-5. doi: 10.1097/MCO.0000000000000228. PMID 26418822
- [Result] Vahia VN. Diagnostic and statistical manual of mental disorders 5: A quick glance. Indian J Psychiatry. 2013 Jul;55(3):220-3. doi: 10.4103/0019-5545.117131. No abstract available. PMID 24082241
- [Result] Kordulewska NK, Kostyra E, Piskorz-Ogorek K, Moszynska M, Cieslinska A, Fiedorowicz E, Jarmolowska B. Serum cytokine levels in children with spectrum autism disorder: Differences in pro- and anti-inflammatory balance. J Neuroimmunol. 2019 Dec 15;337:577066. doi: 10.1016/j.jneuroim.2019.577066. Epub 2019 Sep 15. PMID 31629288
- [Result] Siniscalco D, Schultz S, Brigida AL, Antonucci N. Inflammation and Neuro-Immune Dysregulations in Autism Spectrum Disorders. Pharmaceuticals (Basel). 2018 Jun 4;11(2):56. doi: 10.3390/ph11020056. PMID 29867038